CLINICAL TRIAL: NCT03538067
Title: Influence of Balloon Inflation Techniques and Plaque Characteristics on Stent Under-expansion in Percutaneous RevasculariSaTion (BURST)
Brief Title: Balloon Inflation and Plaque Morphology in Revascularisation (BURST)
Acronym: BURST
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 212423
Record Dates: First submitted 2017-07-31; First posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease; Atherosclerosis
Keywords: percutaneous coronary intervention; stent apposition; stent deployment; stent expansion; intravascular ultrasound
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Paired sample group: Patients with symptomatic coronary artery disease (stable, NSTEACS) undergoing planned percutaneous coronary intervention with intravascular ultrasound (IVUS) guidance
  Interventions: Procedure: Percutaneous coronary intervention (PCI)

INTERVENTIONS:
Procedure: Percutaneous coronary intervention (PCI) — Patients will undergo PCI with intravascular ultrasound (IVUS) as part of standard clinical care in accordance with operator discretion. The research protocol will be observational - using IVUS to determine the effects of balloon inflation time, balloon inflation pressure, balloon type, atherosclerotic plaque morphology on stent expansion (minimal luminal area, MLA)

SUMMARY:
This study will look at the effects of standardised balloon inflation times, pressure and balloon types and atherosclerotic plaque morphology on the procedural results of percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Patients presenting with symptoms of coronary artery disease (e.g. chest pain - angina) are often treated with stents (referred to as percutaneous coronary intervention, PCI). Stents treat the cause of symptoms by improving blood flow to the heart muscle through expanding a narrowed, or diseased segment within a coronary artery. The procedure involves the inflation of a balloon to expand the stent inside the artery. As part of standard clinical care multiple balloon inflations are required during the procedure. Deficiencies in the expansion of the stent at the time of the procedure are associated serious complications such as stent blockages or re-narrowing of the artery, either of which may not occur until much later.

Improvements to the technique of stent expansion are therefore highly desirable to improve outcomes for patients. A number of factors are thought to influence the success of the procedure, including: the type of balloon used to inflate the stent, the pressure used and the duration of balloon inflation. Another important factor may be the mechanical properties of the narrowed segment of the artery (plaque) and how they interact with the stent. At present however, there is no consensus view and the practise of individual cardiologists consequently remains highly variable.

The aim of this study is better characterise relationship between pressure and duration of balloon inflation, type of balloon used and plaque properties during stent procedures using state-of-the-art imaging. Although assessment of each of these factors by a cardiologist is already included as part of standard care, our research protocol will focus the analysis into a systematic framework to allow conclusions to be drawn. The findings will used better inform cardiologists of the technical modifications that can help improve stenting procedures and translate to better outcomes for patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic coronary artery disease (stable angina, non-ST elevation acute coronary syndromes) undergoing percutaneous coronary intervention with intracoronary ultrasound (IVUS) guidance
* Patients > 18 years
* De novo coronary stenoses in native coronary arteries
* Written informed consent

Exclusion Criteria:

* ST-elevation acute coronary syndrome
* Haemodynamic instability
* Cardiogenic shock
* Severe renal dysfunction (eGFR < 30 ml/min/1.73m2)
* In-stent restenosis
* Chronic total occlusions
* Saphenous vein and arterial bypass grafts
* Patients who are currently enrolled in any other study where involvement in this study would involve significant deviation from either protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic coronary artery disease (stable angina, non-ST elevation acute coronary syndromes) already referred for coronary intervention will be prospectively enrolled sequentially as they attend the St Thomas' Cardiac Catheterisation Laboratories.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
In-stent minimal luminal area (MLA, mm2) | Immediate - peri-procedurally
  As measured by intravascular ultrasound

SECONDARY OUTCOMES:
Plaque characteristics | Immediate - peri-procedural
  As determined by virtual histology intravascular ultrasound (VH-IVUS)
Stent deployment | Immediate - peri-procedural
  Determined by intravascular ultrasound (IVUS - MUSIC Criteria)
Peri-procedural myocardial infarction | Immediate - peri-procedural
  In accordance with academic research consortium (ARC) definition

CONTACTS AND LOCATIONS:
Overall Officials: Simon Redwood, MD FRCP FACC, Principal Investigator — King's College London, Guy's and St Thomas' Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided